CLINICAL TRIAL: NCT02749318
Title: Engagement Study: (Multi-site, Practice-Based Research Network (PBRN) Prospective Clinical Trial to Assess if Knowledge of Genetic Risk Changes Behavior)
Brief Title: Dental Engagement Study Behavior Modification
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company Assets Being Sold
Sponsor: Interleukin Genetics, Inc. (Industry)
Collaborators: Duke University (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ILI-16-137-P-US
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: PERIODONTAL DISEASE
Keywords: Behavior Modification; Genetic Testing; Risk Management; Oral Health Care
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Consented patients who complete the initial Experimental Group Questionnaire, receive a prophylaxis, have the IL-1 genetic test for risk of severe periodontitis performed, their dental records monitored for 18 months post-enrollment, and answer a Study Completion Questionnaire 18 months post-enrollment.
  Interventions: Genetic: IL-1 genetic test for risk of severe periodontitis
- Usual Care Group (No Intervention): Consented patients who complete the initial Usual Care Group Questionnaire, receive a prophylaxis and have their dental records monitored for 18 months post-enrollment.

INTERVENTIONS:
Genetic: IL-1 genetic test for risk of severe periodontitis — DNA obtained by cheek swab analyzed for four variations (SNPs) in the IL-1beta gene to determine whether patient is at elevated risk for more severe periodontal disease.
  Other Names: PerioPredict® Genetic Risk Test
  Arms: Experimental Group

SUMMARY:
This is a pilot study to determine whether knowledge gained by an individual of genetic risk for severe periodontitis changes the patient's health behavior as measured by an increased frequency of their preventive dental office visits. In addition to the primary objectives of the study, the overall design and logistics will be used to inform a possible future study.

DETAILED DESCRIPTION:
Data to be analyzed in this study will be gathered through a patient questionnaire, genetic testing and tracking of preventive dental office visits. Eight hundred (800) total participants will be randomly assigned to either the Usual Care or Experimental Groups. Two hundred participants will be assigned to the Usual Care Group and 600 will be assigned to the Experimental Group. It is anticipated that approximately 17% (~100) of the Experimental Group subjects will refuse to enroll in the study, leaving a final total of approximately 500 subject in this group. Within the Experimental Group, 125 subjects positive for the IL-1 genetic test (PerioPredict® Genetic Risk Test, Interleukin Genetics, Inc., Waltham, MA) will be identified and ~375 will test negative for the IL-1 genetic test.

The Sponsor will enter the subject's dental office registration number into a master spreadsheet and randomly assign every fourth patient to the Usual Care Group and all others will be assigned into the Experimental Group. Information about the study and informed consent will be made available by the dental office for the specific groups, either by directing to a website location with videos and ICFs, or alternatively by by dental office showing informational videos on provided tablet and gathering signed hardcopy ICFs at schedule first visit.

ELIGIBILITY:
Inclusion Criteria:

* All adult (18 years of age or older) patients from multi-site, practice-based research network dental offices who have dental insurance coverage for preventive care twice per year, but have only used the benefit once per year in the past 2-3 years.

Exclusion Criteria:

* Patients who previously have had an IL-1 dental genetic test.
* Patients who have been diagnosed with periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The number of preventive oral health care visits per patient (Dental office visit record review) | 18 months from enrollment
  Frequency of preventive oral health care visits within 18 months of enrollment.

SECONDARY OUTCOMES:
Questionnaire on patient demographics and dental healthcare behavior | At enrollment by survey
  Reasons for not fully utilizing preventive oral health care insurance benefits
Questionnaire on changes in oral health care behavior and attitudes on genetic testing | 18 months after enrollment
  Reasons for changes in frequency of preventive oral health care behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth S Kornman, D.D.S. PhD., Principal Investigator — Interleukin Genetics, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu X, Offenbacher S, Lomicronpez NJ, Chen D, Wang HY, Rogus J, Zhou J, Beck J, Jiang S, Bao X, Wilkins L, Doucette-Stamm L, Kornman K. Association of interleukin-1 gene variations with moderate to severe chronic periodontitis in multiple ethnicities. J Periodontal Res. 2015 Feb;50(1):52-61. doi: 10.1111/jre.12181. Epub 2014 Apr 2. PMID 24690098
- [Background] Giannobile WV, Braun TM, Caplis AK, Doucette-Stamm L, Duff GW, Kornman KS. Patient stratification for preventive care in dentistry. J Dent Res. 2013 Aug;92(8):694-701. doi: 10.1177/0022034513492336. Epub 2013 Jun 10. PMID 23752171